CLINICAL TRIAL: NCT01701778
Title: Double-blind Randomized Controlled Trial of Caudal Versus Intravenous Dexmedetomidine for Supplementation of Caudal Analgesia in Children
Brief Title: Caudal Versus Intravenous Dexmedetomidine for Supplementation of Caudal Analgesia in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yao Yusheng (Other)
Collaborators: West China Hospital (Other)
Responsible Party: Sponsor-Investigator, Yao Yusheng, Double-blind randomized controlled trial of caudal versus intravenous dexmedetomidine for supplementation of caudal analgesia in children, Fujian Provincial Hospital
Organization: Fujian Provincial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FujianPH; FujianPH-TRC-121002 (Registry Identifier: Fujian Provicial Hospital)
Record Dates: First submitted 2012-10-02; First posted 2012-10-05 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Inguinal Hernia; Cryptorchidism
Keywords: Dexmedetomidine; Postoperative pain reaction; anesthesia; children
MeSH Terms: conditions — Hernia, Inguinal; Cryptorchidism | interventions — Dexmedetomidine; Levobupivacaine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Caudal Dexmedetomidine (Experimental): Caudal: Levobupivacaine 0.25% 1ml/kg and dexmedetomidine 1µg/kg
  Intravenous: 10 ml normal saline
  Anesthesia was induced and maintained with sevoflurane
  Interventions: Drug: Caudal Dexmedetomidine; Drug: sevoflurane
- Intravenous Dexmedetomidine (Experimental): Caudal: Levobupivacaine 0.25% 1ml/kg
  Intravenous: dexmedetomidine 1µg/kg
  Anesthesia was induced and maintained with sevoflurane
  Interventions: Drug: Intravenous Dexmedetomidine; Drug: sevoflurane
- Placebo (Placebo Comparator): Caudal: Levobupivacaine 0.25% 1ml/kg
  Intravenous: 10 ml normal saline
  Anesthesia was induced and maintained with sevoflurane
  Interventions: Drug: Placebo; Drug: sevoflurane

INTERVENTIONS:
Drug: Caudal Dexmedetomidine — Caudal: Levobupivacaine 0.25% 1ml/kg and dexmedetomidine 1µg/kg
  Intravenous: 10 ml normal saline
  Other Names: Precedex
  Arms: Caudal Dexmedetomidine
Drug: Intravenous Dexmedetomidine — Caudal: Levobupivacaine 0.25% 1ml/kg
  Intravenous: dexmedetomidine 1µg/kg
  Other Names: Precedex
  Arms: Intravenous Dexmedetomidine
Drug: Placebo — Caudal: Levobupivacaine 0.25% 1ml/kg
  Intravenous: 10 ml normal saline
  Other Names: Levobupivacaine
  Arms: Placebo
Drug: sevoflurane — Induction and maintain anaesthesia

SUMMARY:
The purpose of this study is to compare the effects of caudal dexmedetomidine with intravenous dexmedetomidine on caudal levobupivacaine analgesia in children undergoing lower abdominal surgeries.

DETAILED DESCRIPTION:
Single shot caudal epidural block is one of the most widespread technique for pediatric pain management after infraumbilical surgical procedures.However, in a significant proportion of patients, despite good initial analgesia from a caudal block with local anesthetic, pain develops after the block resolves.

Dexmedetomidine is used increasingly in pediatric anesthesia practice to prolong the duration of action of caudal block with a local anesthetic agent.But which route of administration of clonidine is the most beneficial remains unknown.

The investigators performed prospective randomized double-blind study to compare the effects of caudal dexmedetomidine with intravenous dexmedetomidine on postoperative analgesia after caudal levobupivacaine for inguinal herniorrhaphy or orchidopexy surgery.

90 children (ASAⅠorⅡ,aged 2-5 yr) undergoing unilateral orchiopexy or inguinal herniorrhaphy were included in this study. Anesthesia was induced with sevoflurane via a facemask, followed by placement of a laryngeal mask airway. Anesthesia was maintained with sevoflurane 2-3% in oxygen-air.Then,caudal block was applied. Patients were randomly assigned in three groups. Group Cau-DEX (n = 30): Caudal Levobupivacaine 0.25% 1ml/kg plus dexmedetomidine 1µg/kg and 10 ml normal saline i.v.;Group IV-DEX(n = 30): Levobupivacaine 0.25% 1ml/kg and dexmedetomidine 1µg/kg(10 ml)i.v.;Group Placebo(n = 30): Levobupivacaine 0.25% and 10 ml normal saline intravenous.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II
* aged 2-5 yr
* Undergoing unilateral orchiopexy/inguinal hernia repair

Exclusion Criteria:

* Hypersensitivity to any local anesthetics
* Patient has history of allergy, intolerance, or reaction to dexmedetomidine
* Infections at puncture sites
* Bleeding diathesis
* Preexisting neurological disease
* Diabetes mellitus
* Children with uncorrected cardiac lesions
* Children with heart block or liver impairment

Ages: 2 Years to 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Time to first rescue medication | From the administration of the caudal block to the first registration of a CHIPPS scores≥4,assessed up to 24h
  the Children and Infants Postoperative Pain Scale (CHIPPS)

SECONDARY OUTCOMES:
the number of patients not requiring rescue analgesia | After surgery,up to 24h
  the quality of postoperative pain control
the sedation score | After surgery, every 15min for the first 2 h, every 30min for the next 2h, hourly for the next 4h
  sedation was assessed using the Modified Ramsay Sedation Score
Residual motor block | After awake,participants will be followed every 30min for the first 2h, hourly for the next 4h
  the degree of motor blockade was assessed using a modified Bromage scale
the incidence of emergence agitation | Participants will be followed for the duration of PACU stay, an expected average of 2 hours
  The incidence of emergence agitation was evaluated by the Pediatric Anesthesia Emergence Delirium Scale(PAED)
side effects | From the administration of the caudal block until the end of study period, assessed up to postoperative 24h
  side effects including bradycardia, hypotension, hypoxemia, nausea, vomiting and urinary retention
Pain intensity | after surgery, 30min for first 4h, hourly for the next 4h and thereafter every 2h,assessed up to 24h
  Participants will be assessed with Children and Infants Postoperative Pain Scale (CHIPPS)

CONTACTS AND LOCATIONS:
Overall Officials: Yusheng Yao, M.D., Principal Investigator — Fujian Provincial Hospital; Yanqing Chen, M.D., Principal Investigator — Fujian Provicial Hospital; Jin Liu, M.D., Study Director — West China Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

REFERENCES:
- [Derived] Yao Y, Yu C, Zhang X, Guo Y, Zheng X. Caudal and intravenous dexmedetomidine similarly prolong the duration of caudal analgesia in children: A randomized controlled trial. Paediatr Anaesth. 2018 Oct;28(10):888-896. doi: 10.1111/pan.13469. PMID 30302881